CLINICAL TRIAL: NCT00964314
Title: Prospective Study With RCT Designed for Evaluation of TCM Five Elements Music Therapy Improving Quality of Life in Patients With Advanced Cancer
Brief Title: Traditional Chinese Medicine Five Elements Music Therapy Improving Quality of Life in Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Liao Juan, Oncology Department of Xi Yuan Hospital, China Academy of Chinese Medicine Sciences, Ministry of Science and Technology of the People´s Republic of China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WJB720603
Record Dates: First submitted 2009-08-19; First posted 2009-08-24 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Cancer
Keywords: advanced cancer; TCM five elements music therapy; quality of life (QOL)
MeSH Terms: conditions — Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- five elements music (Experimental): Listening TCM five elements music therapy（TCMMT）based on conventional therapy in China.
  Interventions: Other: music
- western music (Active Comparator): Listening western music based on conventional therapy in China.
  Interventions: Other: music
- Without music (No Intervention): no music therapy will be done in the arm.
  Interventions: Other: music

INTERVENTIONS:
Other: music — Experimental Group one : Listening TCM five elements music therapy（TCMMT）based on conventional therapy in China.
  Experimental Group two: Listening western music based on conventional therapy in China.
  Control Group: no music therapy will be done.

SUMMARY:
The study objective is to evaluate the effectiveness of Traditional Chinese Medicine (TCM) five elements music therapy improving quality of life for patients with advanced cancer, as well as establishing the standard operating procedures (SOP) for it.

DETAILED DESCRIPTION:
Design: As randomized controlled trial (RCT) with un-blinded design will be done.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participation will be enrolled based on diagnostic criteria.
* Advanced cancer patient with more than 50 scores of Karnofsky Performance Score (KPS).
* Diagnosis of advanced cancer
* Patients who are willing to be subject with taking part in this research voluntarily.
* No prior experience with TCM music therapy.
* Newly admitted to TCM oncology department for 3 weeks treatment course.

Exclusion Criteria:

* Complicated diagnose or one who don't consistent with inclusion criteria.
* Patients suffering from psychosis or diagnosis, or psychiatric diagnoses (e.g., schizophrenia).
* Suffering from acute organ prostration or other condition of demanding to rescue，inability for accepting music therapy.
* One don't read or fill in diary owing to some causes, such as state of the art or acuity of vision
* One suffering from hearing disturbance
* Accepted TCM five elements music therapy in the past.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Comparison of KPS Qol, and Diary at baseline and endpoint in each group (data for < 70 year old group). | Difference of(pro-post)treatment for KPS,Qol, Diary
  Comparison of Qol, KPS, Diary at baseline and endpoint, the result shown here were significantly different for all terms in TCM five elements music group, p=0. p=0.0015, p=0.0015 respectively. However, no significant difference was seen for all terms in Western music group and the no music group respectively (See Table 3).
Comparison of KPS Qol, and Diary at baseline and endpoint in each group (data for the >70 year old group). | Difference of(pro-post)treatment for KPS,Qol, Diary
  Comparison of Qol, KPS and Diary score at baseline and endpoint results show there was a significant difference for the QoL in TCM five elements music group, p value is 0.0062. However, there was no significant difference for the KPS and Diary score in each group respectively(See Table 4).

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yu fei, doctor, Study Director — Oncology department of Xi Yuan Hospital, China Academy of Chinese Medical Sciences
Locations (2):
- China (2):
  - Xi-Yuan Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Oncology Department of Xi Yuan hospital, Beijing, HaiDian District

REFERENCES:
- See also: Related Info — http://www.cctcm.com